CLINICAL TRIAL: NCT03857230
Title: Study of Safety, Tolerance and Pharmacokinetics of Primapur and Gonal-f Upon Single-dose Subcutaneous Administration in Healthy Volunteers
Brief Title: The Safety and Pharmacokinetics of Primapur and Gonal-f
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IVFarma LLC (Industry)
Collaborators: NADIM LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FSG-01-01
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Area Under Curve; Pharmacokinetics; Absorption
Keywords: follitropin alfa; follicle stimulating hormone; hormones, hormone substitutes, and hormone antagonists; physiological effects of drugs; biosimilar; bioequivalence
MeSH Terms: interventions — follitropin alfa; Glycoprotein Hormones, alpha Subunit; Follicle Stimulating Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A: Primapur - Gonal-F (Experimental): Subjects were randomly assigned to receive treatment sequence A: single subcutaneous injection of 300 IU Primapur on study day 1, after 10 days of wash out period a single subcutaneous injection of 300 IU Gonal-F.
  Interventions: Drug: Follitropin alfa (Primapur); Drug: Follitropin alfa (Gonal-F)
- Sequence B: Gonal-F - Primapur (Active Comparator): Subjects were randomly assigned to receive treatment sequence B: single subcutaneous injection of 300 IU Gonal-F on study day 1, after 10 days of wash out period a single subcutaneous injection of 300 IU Primapur.
  Interventions: Drug: Follitropin alfa (Primapur); Drug: Follitropin alfa (Gonal-F)

INTERVENTIONS:
Drug: Follitropin alfa (Primapur) — During the crossover pharmacokinetic phase, after 42 days of combined oral contraceptive (ethinylestradiol and drospirenone) administration subjects with endogenous level of follicle stimulating hormone (FSH) less than 5 IU/l were randomly assigned to receive one of the following treatment sequences:
  Sequence A: Single subcutaneous injection of 300 IU Primapur on study day 1, after 10 days of wash out a single subcutaneous injection of 300 IU Gonal-F.
  Sequence B: Single subcutaneous injection of 300 IU US Gonal-F on study day 1, after 10 days of wash out a single subcutaneous injection of 300 IU Primapur.
  Other Names: Follitropin alpha; Follitropin
Drug: Follitropin alfa (Gonal-F) — During the crossover pharmacokinetic phase, after 42 days of combined oral contraceptive (ethinylestradiol and drospirenone) administration subjects with endogenous level of follicle stimulating hormone (FSH) less than 5 IU/l were randomly assigned to receive one of the following treatment sequences:
  Sequence A: Single subcutaneous injection of 300 IU Primapur on study day 1, after 10 days of wash out a single subcutaneous injection of 300 IU Gonal-F.
  Sequence B: Single subcutaneous injection of 300 IU US Gonal-F on study day 1, after 10 days of wash out a single subcutaneous injection of 300 IU Primapur.
  Other Names: Follitropin alpha; Follitropin

SUMMARY:
The purpose of the current phase I study was to establish bioequivalence, safety, and tolerance of single 300 IU subcutaneous dose of follitropin alfa biosimilar (Primapur) in comparison to that of reference follitropin alfa preparation (Gonal-F) in healthy young female volunteers.

DETAILED DESCRIPTION:
A Phase I, prospective, randomized, open-label, crossover, 2-period, two treatment, clinical study in healthy female volunteers.

Objectives of the study:

1. To evaluate the frequency and severity of adverse events (AE) following a single 300 IU subcutaneous injection of Primapur (IVFarma, LLC, Russia) and Gonal-F (Merck Serono S.p.A., Italy) to healthy volunteers.
2. To determine the AUC0-t value of Primapur following a single 300 IU subcutaneous injection to healthy volunteers.
3. To determine the T½ value of Primapur following a single 300 IU subcutaneous injection to healthy volunteers.
4. To determine the Сmax value of Primapur following a single 300 IU subcutaneous injection to healthy volunteers.
5. To determine the Tmax value of Primapur following a single 300 IU subcutaneous injection to healthy volunteers.
6. To compare the obtained pharmacokinetic characteristics of Primapur and Gonal-F.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female volunteers aged 18 to 40 years.
2. Body mass index (BMI) of 18.5 to 30.0 kg/m2.
3. Subjects who have used oral contraceptives for at least 2 menstrual cycles before study entry.
4. Regular menstruation cycle (24 to 35 days) before initiation of oral contraception.
5. Presence of both ovaries.
6. Subjects who are negative for drugs of abuse and alcohol tests at screening.
7. Subjects who are healthy as validated by pre study medical history, physical examination.
8. Subjects with acceptable clinical laboratory test results.
9. A signed informed consent form that confirms in writing the volunteer's consent to participate in this clinical study and the volunteer's willingness to comply with all physician recommendations and protocol limitations for the time of participation in the clinical study.
10. Ability to comply with the requirements of the protocol.
11. Participants in the study, as well as their sexual partners, are knowledgeable and willing to voluntarily, starting from the week before being included in the study and up to 4 weeks after the last dose of the study drug, and in addition to the contraceptive used, use at least 1 barrier contraceptive method or spermicide.

Exclusion Criteria:

1. Hypersensitivity to follitropin alpha, combined oral contraceptive (ethinylestradiol and drospirenone) or excipients.
2. Allergy, angioedema (hereditary or idiopathic) in history.
3. Previous history of ovarian hyperstimulation syndrome (OHSS).
4. Inability to establish a venous catheter for blood sampling.
5. Presence of polycystic ovaries (PCO) and ovarian cysts.
6. Neoplasia and a history of malignant disease.
7. Deep vein thrombosis, pulmonary embolism.
8. Subjects with impaired thyroid function.
9. Regular usage or administration of any drugs, including non-prescription drugs, vitamins, homeopathic remedies and dietary supplements, less than 2 weeks before the study (with the exception of contraceptive pills).
10. Admission less than 2 months before the start of the study of drugs that have a pronounced effect on hemodynamics, liver function, and medication contained follicle stimulating hormone (FSH), luteinizing hormone (LH), chorionic gonadotropin (hCG), clomiphene, gonadotropin-releasing hormone (GnRH) analogues.
11. Cardiovascular, bronchopulmonary, nervous, endocrine systems, gastrointestinal tract, liver, kidney, hematopoietic, immune systems, mental diseases.
12. Acute infectious diseases less than 4 weeks before the start of the study.
13. Systolic pressure less than 100 mm or above 130 mm Hg; diastolic pressure less than 70 mm or above 90 mm Hg; heart rate less than 60 or more than 80 beats/min.
14. Blood donation less than 3 months before the start of the study.
15. Participation in clinical studies of drugs less than 3 months before the start of the present study.
16. More than 5 alcohol units per week (1 unit is equal to 50 ml of a strong alcoholic drink, 200 ml of dry wine or 500 ml of beer) or anamnestic information about alcoholism, drug addiction, drug abuse.
17. Smoking more than 5 cigarettes/day.
18. Narcomania, alcoholism.
19. Presence of pregnancy.
20. Lactating.
21. Any reason that, in the opinion of the investigator, could interfere with safety of the subject or interfere with the objectives of the study.
22. Subjects with a lactose intolerance, lactase deficiency or glucose-galactose malabsorption.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan G Gordeev, D.Sc., MD, Principal Investigator — O.M. Filatov Municipal Clinical Hospital N 15
Locations (1):
- O.M. Filatov Municipal Clinical Hospital N 15, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tyul'kina EE, Gordeev IG, Grebenkin DYu, Kazei VA, Tsikarishvili MM, Luchinkina EE, et al. Randomized crossover comparative study of safety, tolerance and pharmacokinetics of Primapur vs. Gonal-f upon single-dose subcutaneous administration in healthy volunteers. Eksperimental'naya i Klinicheskaya Farmakologiya. 2017; 80(4): 13-17 (in Russian).
- See also: Link to a publisher site with a full-text article — https://doi.org/10.30906/0869-2092-2017-80-4-13-17

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Duration of participation was about 73 days: screening period (up to 7 days), preparation period (up to 28 days), the 1st period (9 days), the 2nd period (9 days), and the follow-up period (28 days starting from the first day of the 2nd period). The wash-out period is 10 days.
Pre-assignment Details: 28 healthy female volunteers aged 18 to 40 years inclusively have been enrolled according to the inclusion and non-inclusion criteria, among them 4 back-ups enrolled in the study to replace the volunteers excluded before the study completion.
Period: Period 1 (Primapur-Gonal-F)
Arm/Group | Sequence A: Primapur - Gonal-F | Sequence B: Gonal-F - Primapur
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Period 2 (Gonal-F-Primapur)
Arm/Group | Sequence A: Primapur - Gonal-F | Sequence B: Gonal-F - Primapur
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Women aged 18 to 40 years; body mass index (BMI) of 18.5 to 30 kg/m2
Groups:
- Sequence A: Primapur - Gonal-F: Subjects were randomly assigned to receive treatment sequence A: single subcutaneous injection of 300 IU Primapur on study day 1, after 10 days of wash out a single subcutaneous injection of 300 IU Gonal-F.
- Sequence B: Gonal-F - Primapur: Subjects were randomly assigned to receive treatment sequence B: single subcutaneous injection of 300 IU Gonal-F on study day 1, after 10 days of wash out a single subcutaneous injection of 300 IU Primapur.
- Total: Total of all reporting groups
Arm/Group | Sequence A: Primapur - Gonal-F | Sequence B: Gonal-F - Primapur | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  Periods 1 and 2: <=18 years | 0 | 0 | 0
  Periods 1 and 2: Between 18 and 65 years | 12 | 12 | 24
  Periods 1 and 2: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.92 (4.27) | 26.58 (3.12) | 28.25 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 12 | 12 | 24
Body mass index (BMI) [Mean (Standard Deviation); unit: kg per m2] | 23.41 (3.53) | 22.41 (2.80) | 22.91 (3.16)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration of Follicle Stimulating Hormone (FSH) - Time Curve (AUC(0-192))
Description: Area under curve (AUC), Time frame: From 0 (predose), 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 120, 168 and 192 hours postdose.
  Blood samples to study the pharmacokinetics are to be collected via a venous catheter, which is placed by means of vein puncture before any injection of r-hFSH. Blood sampling were carried out at certain time points according to the specified scheme: - 20 minutes (20 minutes before the drug injection), 0 hours (immediately prior to injection), and 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 120, 168, and 192 hours after each injection of the drug product.
Time Frame: 0-192 hours
Population: Blood sampling were carried out at certain time points according to the specified scheme: - 20 minutes (20 minutes before the drug injection), 0 hours (immediately prior to injection), and 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 120, 168, and 192 hours after each injection of the drug product.
Measure: Geometric Mean (Standard Deviation); unit: mIU*h/ml
Groups:
- Primapur: All subjects who received a single subcutaneous injection of 300 IU Primapur.
- Gonal-F: All subjects who received a single subcutaneous injection of 300 IU Gonal-F.
Arm/Group | Primapur | Gonal-F
Number analyzed (Participants) | 24 | 24
mIU*h/ml | 1202.85 (466.28) | 1241.01 (418.61)
Statistical Analysis 1: Comparison: Primapur vs Gonal-F; Statistical comparison of the obtained results comprised the calculation of parametric bilateral 90 % CIs for the ratios of the corresponding mean values of the pharmacokinetic parameters of the study and comparator drug. The equivalence of the pharmacokinetics of the drug products will be proven if the limits of the evaluated CIs for the ratios of the mean values are in the range of 80.00-125.00%; Test type: Equivalence — The 90% CIs of the ratios of geometric means of log-transformed baseline AUC0-192 were used to assess bioequivalence between Primapur and Gonal-F (bioequivalence range of 80.00% to 125.00%); p = 0.05, ANOVA; Geometric Mean Ratio (%) = 93.31, 90% CI 2-sided [87.25 to 99.79]

2. Primary Outcome: Maximum Serum Concentration of Follicle Stimulating Hormone (FSH) (Cmax)
Description: Maximum serum concentration (Cmax), Time frame: From 0 (predose), 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 120, 168 and 192 hours postdose.
Time Frame: 0-192 hours
Measure: Geometric Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Primapur | Gonal-F
Number analyzed (Participants) | 24 | 24
mIU/ml | 14.32 (4.72) | 16.00 (4.88)
Statistical Analysis 1: Comparison: Primapur vs Gonal-F; Test type: Equivalence — The 90% CIs of the ratios of geometric means of log-transformed baseline Cmax were used to assess bioequivalence between Primapur and Gonal-F (bioequivalence range of 80.00% to 125.00%); p = 0.05, ANOVA; Geometric Mean Ratio (%) = 87.93, 90% CI 2-sided [82.85 to 93.33]

3. Secondary Outcome: Time to Reach a Maximum Follicle Stimulating Hormone (FSH) Serum Concentration (Tmax)
Description: Time to reach a maximum serum concentration (Tmax), Time frame: From 0 (predose), 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 120, 168 and 192 hours postdose.
Time Frame: 0-192 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Primapur | Gonal-F
Number analyzed (Participants) | 24 | 24
hours | 18.70 (5.77) | 19.22 (4.93)

4. Secondary Outcome: Follicle Stimulating Hormone (FSH) Apparent Terminal Half-life (T1/2)
Description: Terminal half-life (T1/2), Time frame: From 0 (predose), 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 120, 168 and 192 hours postdose.
Time Frame: 0-192 hours
Measure: Geometric Least Squares Mean (Standard Deviation); unit: hours
Arm/Group | Primapur | Gonal-F
Number analyzed (Participants) | 24 | 24
hours | 70.78 (32.54) | 71.71 (33.47)

5. Other Pre Specified Outcome: Elimination Rate Constant (Kel)
Description: Elimination rate constant (Kel): Time frame: From 0 (predose), 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 120, 168 and 192 hours postdose.
Time Frame: 0-192 hours
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Primapur | Gonal-F
Number analyzed (Participants) | 24 | 24
1/h | 0.01 (0.003) | 0.01 (0.006)

ADVERSE EVENTS:
Time Frame: From the study day 1 to day 56.
Description: An adverse event was defined as any adverse event that began following the first dose of follitropin alfa administration till the end of follow-up period. Adverse events were reported from the 1st period (9 days), wash out period (10 days), 2nd period (9 days) and follow-up period (28 days).
Arm/Group | Primapur | Gonal-F
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 11/24 | 10/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primapur (N=24) | Gonal-F (N=24)
Laboratory investigations (Investigations) | 8 (11) | 8 (11)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT03857230/Prot_SAP_000.pdf